CLINICAL TRIAL: NCT05020262
Title: A Retrospective, Single-center, Readerblind, Nonrandomized Clinical Trial Was Conducted to Evaluate the Function of Incisive CT Precise Image and Precise Cardiac Function
Brief Title: Incisive CT Clinica Trial Protocol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Collaborators: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PD_CT_Incisive CT_2021_11264
Record Dates: First submitted 2021-08-10; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: CT Images

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Test Group: Using PI/PC reconstruct raw data
  Interventions: Other: CT Image reconstruction
- Control Group: Using Idose4/Cardiac Image reconstruct raw data
  Interventions: Other: CT Image reconstruction

INTERVENTIONS:
Other: CT Image reconstruction — Retrospectively collects CT Images and reconstruct using PI/PC and Idose4/Cardiac Images to assessment the performance of the two new software functions of Incisive CT. No direct intervention to patients. And ICF is exempted by EC.

SUMMARY:
The purpose of this study was to evaluate whether the new features of Incisive CT: Precise Image, (PI) and Precise Cardiac (PC) had the expected effectiveness

ELIGIBILITY:
Inclusion Criteria:

* The original data of the images are from the patient base in the age range of 18 to 75 years (18≤ age ≤75 years)
* Original image data are collected in Incisive CT (version 4.5) and traceable;
* Time range for inclusion of original image data: from the start of the clinical trial to the completion of collection in compliance with this protocol;

Exclusion Criteria:

- The investigator deemed it inappropriate to include the original image data for this clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The original data of the images are from the patient base in the age range of 18 to 75 years (18≤ age ≤75 years)
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The quality of PI/PC and iDose4/ cardiac imaging reconstructed images was basically equal or above 3 score | through study completion, an average of 2months
  Scoring criteria 5 points The image quality of PI/PC is better than that of iDose4/ cardiac imaging, which can be used for diagnosis, very satisfied 4 points The image quality of PI/PC is better than that of contrast products, and the image of iDose4/ cardiac imaging can be used for diagnosis, satisfactory 3 points The image quality of PI/PC is basically equivalent to that of iDose4/ cardiac imaging. The image quality is defective, which does not affect the diagnosis, but is normal 2. The image quality of PI/PC is not lower than iDose4/ cardiac imaging, but the image quality is poor, which affects the diagnosis and is not satisfactory
  1 points The image quality is lower than iDose4/ cardiac imaging after using PI/PC, the image quality is poor, cannot diagnose, unsatisfactory

SECONDARY OUTCOMES:
Imaging reconstruction enhancement condition using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score enhancement 5 points - Very satisfied very clear and good, can be used for diagnosis 4 points - Satisfaction is clear and good and can be used for diagnosis 3 points - Generally defective, acceptable, without affecting diagnosis 2 points - Unsatisfactory enhancement is poor, affecting diagnosis
  1 point - Unsatisfactory enhancement is poor and cannot be diagnosed
Imaging reconstruction diagnostic confidence using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score diagnostic confidence 5 points - Very satisfied the lesion or tissue structure is shown very clearly and can be used for diagnosis Score 4 - Satisfied that the lesion or tissue structure is clearly displayed and can be used for diagnosis 3 points - Generally the lesion or tissue structure is shown with acceptable clarity and does not affect the diagnosis 2 points - unsatisfactory lesion or tissue structure showing poorly, affecting diagnosis
  1 point - Unsatisfactory lesion or tissue structure is not clearly displayed and cannot be diagnosed
Imaging reconstruction clarity using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score clarity 5 points - Very satisfied with the clear edge, the details show very clear and clear and can be used for diagnosis 4 points - Satisfied with a clear edge, showing clear and clear details that can be used for diagnosis 3 points - General clarity acceptable without prejudice to diagnosis 2 points - Undersatisfied edges and details show smooth, unclear, affecting diagnosis
  1 point - Unsatisfied edges and detail display that is too smooth and unclear to affect diagnosis
Imaging reconstruction Noise level using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score noise level 5 points - Very satisfied with very low or no noise, can be used for diagnosis 4 points - Satisfied with low or mild noise, can be used for diagnosis 3 points - General The noise value is normal, acceptable and does not affect the diagnosis 2 points - unsatisfactory high noise, affecting diagnosis
  1 point - Dissatisfaction with high noise and excessive noise that affects diagnosis
Imaging reconstruction Image texture using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score image texture 5 points - Very satisfied with texture very clear, intuitive feel similar to high dose scan image quality, can be used for diagnosis 4 points - Satisfied with clear texture and good image quality for diagnostic purposes 3 points - General texture is normal, image edges or some areas of speckled blur or smoothness, but acceptable, does not affect the diagnosis Score 2 - An undersatisfied image has acceptable speckled blurring that will not be misdiagnosed as lesions and affect the diagnosis
  1 point - Unsatisfactory image texture and poor texture, blotchy, affecting diagnosis
Imaging reconstruction Image artifacts using PI/PC compared with using iDose4/ cardiac basically equivalence to or above 3 score | through study completion, an average of 2months
  Score image artifacts 5 points - Very satisfied no artifacts, can be used for diagnosis 4 points - Satisfied with few artifacts, can be used for diagnosis 3 points - Generally acceptable artifacts that do not affect diagnosis 2 points - undersatisfaction has some artifacts that affect diagnosis
  1 point - Unsatisfied with severe artifacts that affect diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Chao Du, Deputy Director, Principal Investigator — The Second Hospital of Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No